CLINICAL TRIAL: NCT06929962
Title: Vonoprazan-Amoxicillin Dual Sequential Therapy For Helicobacter Pylori-infected Treatment-naive Patients：A Randomized, Open-label, Parallel-controlled , Multicenter Clinical Trial
Brief Title: VA Dual Sequential Therapy
Acronym: JSHERO3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Ye, Associate professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025JSHERO3
Record Dates: First submitted 2025-03-26; First posted 2025-04-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Vonoprazan; Amoxicillin; Sequential therapy; Eradication
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 14-day Vonoprazan-Amoxicillin dual sequential therapy (Experimental): First 7 days (Day 1 to Day 7): 20mg Vonoprazan twice times daily and 1g Amoxicillin twice times daily; Last 7 days (Day 8 to Day 14): 20mg Vonoprazan twice times daily and 1g Amoxicillin three times daily.
  Interventions: Drug: Vonoprazan and Amoxicillin for the first 7 days; Drug: Vonoprazan and Amoxicillin for the second 7 days
- 10-day Vonoprazan-Amoxicillin dual sequential therapy (Experimental): First 5 days (Day 1 to Day 5): 20mg Vonoprazan twice times daily and 1g Amoxicillin twice times daily; Last 5 days (Day 6 to Day 10): 20mg Vonoprazan twice times daily and 1g Amoxicillin three times daily.
  Interventions: Drug: Vonoprazan and Amoxicillin for the first 5 days; Drug: Vonoprazan and Amoxicillin for the second 5 days
- 14-day Vonoprazan-Amoxicillin dual therapy (Active Comparator): 20mg Vonoprazan twice times daily and 1g Amoxicillin three times daily for 14 days.
  Interventions: Drug: Vonoprazan and Amoxicillin for 14 days

INTERVENTIONS:
Drug: Vonoprazan and Amoxicillin for the first 7 days — 20mg Vonoprazan twice times daily and 1g Amoxicillin twice times daily for 7 days
  Other Names: L-VA-7
  Arms: 14-day Vonoprazan-Amoxicillin dual sequential therapy
Drug: Vonoprazan and Amoxicillin for the first 5 days — 20mg Vonoprazan twice times daily and 1g Amoxicillin twice times daily for 5 days
  Other Names: L-VA-5
  Arms: 10-day Vonoprazan-Amoxicillin dual sequential therapy
Drug: Vonoprazan and Amoxicillin for the second 7 days — 20mg Vonoprazan twice times daily and 1g Amoxicillin three times daily for 7 days
  Other Names: H-VA-7
  Arms: 14-day Vonoprazan-Amoxicillin dual sequential therapy
Drug: Vonoprazan and Amoxicillin for the second 5 days — 20mg Vonoprazan twice times daily and 1g Amoxicillin three times daily for 5 days
  Other Names: H-VA-5
  Arms: 10-day Vonoprazan-Amoxicillin dual sequential therapy
Drug: Vonoprazan and Amoxicillin for 14 days — 20mg Vonoprazan twice times daily and 1g Amoxicillin three times daily for 14 days
  Other Names: VADT-14
  Arms: 14-day Vonoprazan-Amoxicillin dual therapy

SUMMARY:
Sequential therapy for Hp was first introduced by Zullo et al. in 2000 and consists of two phases: the first phase involves proton pump inhibitors with one antibiotic, and the second phase involves proton pump inhibitors with two antibiotics. Based on this, the investigators propose a modified sequential therapy, where the first phase uses vonoprazan combined with amoxicillin, and the second phase increases the amoxicillin dosage, forming a high-dose amoxicillin regimen. This new treatment strategy combines the staged nature of sequential therapy with the advantages of high-dose dual therapy, gradually increasing the drug dosage to help patients adapt and reduce side effects (such as nausea, vomiting, and diarrhea), thereby improving patient tolerance.

The primary aim of this study is to compare the vonoprazan combined with high-dose amoxicillin sequential therapy with standard dual therapy (14-day regimen) in terms of Hp eradication rates, efficacy, side effect incidence, and patient compliance, to evaluate its improved effectiveness. Additionally, the study will explore the impact of a shortened treatment duration on the modified dual sequential therapy's efficacy for Hp infection.

Eligible participants in this study will be randomly assigned to one of the following three treatment groups based on a pre-generated randomization sequence:

Control Group: Vonoprazan combined with high-dose amoxicillin dual therapy for 14 days (VADT-14): Vonoprazan 20mg twice daily + Amoxicillin 1g three times daily.

Experimental Group 1: Vonoprazan combined with amoxicillin dual sequential therapy for 14 days (VAST-14):

Days 1 to 7: Vonoprazan 20mg twice daily + Amoxicillin 1g twice daily. Days 8 to 14: Vonoprazan 20mg twice daily + Amoxicillin 1g three times daily.

Experimental Group 2: Vonoprazan combined with amoxicillin dual sequential therapy for 10 days (VAST-10):

Days 1 to 5: Vonoprazan 20mg twice daily + Amoxicillin 1g twice daily. Days 6 to 10: Vonoprazan 20mg twice daily + Amoxicillin 1g three times daily.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) is a Gram-negative, spiral-shaped, microaerophilic bacterium that colonizes the gastric mucosa. HP infection is a key pathogenic factor for peptic ulcers and chronic active gastritis and is closely associated with the development of gastric cancer and mucosa-associated lymphoid tissue lymphoma. Eradicating HP can effectively control disease progression and reduce the risk of related diseases. However, the increasing global antibiotic resistance poses significant challenges to HP eradication, necessitating further exploration of treatment regimens.

Dual therapy was first proposed in the late 1980s for treating HP infection. Given the pH-dependent and time-dependent antibacterial effects of amoxicillin on HP, recent improvements to dual therapy have focused on increasing drug dosage and administration frequency. A 2019 randomized controlled trial in China, including 232 patients, found that the modified dual therapy achieved similar eradication rates to bismuth quadruple therapy but with lower incidence of side effects and treatment costs. The 2022 Chinese guidelines for HP infection treatment recommend bismuth quadruple therapy and high-dose amoxicillin combined with proton pump inhibitors (PPI) as first-line eradication regimens.

Vonoprazan, a novel potassium-competitive acid blocker, offers stronger and more sustained gastric acid suppression compared to traditional PPIs, enhancing the bactericidal effect of amoxicillin. Therefore, vonoprazan is considered a superior choice for dual therapy. A Chinese study showed that a 14-day regimen of vonoprazan (20mg bid) combined with amoxicillin (1.0g tid) achieved similar efficacy and safety to esomeprazole (20mg qid) combined with amoxicillin (750mg qid) (ITT eradication rates: 89% vs. 87.7%, PP eradication rates: 94.1% vs. 92.8%), suggesting it as a potential first-line therapy for HP infection. The 2024 ACG guidelines for HP infection treatment recommend vonoprazan-based dual therapy (20mg bid + 1g tid of amoxicillin for 14 days) as a first-line option.

Sequential therapy for HP infection was first proposed by Zullo et al. in 2000, comprising two phases: the first phase involves 5-7 days of PPI combined with one antibiotic, and the second phase involves 5-7 days of PPI combined with two antibiotics. Studies have shown that the ITT eradication rate for the traditional 14-day sequential therapy regimen is 90.7%, while the 10-day regimen shows a rate of 87.0%. Building on the traditional sequential therapy, the investigators propose a modified sequential therapy strategy. In the first phase, vonoprazan is combined with amoxicillin (1g bid), and in the second phase, the amoxicillin dosage is increased to 1g tid. The proposed regimen is as follows: Days 1-7, vonoprazan (20mg bid) + amoxicillin (1g bid); Days 8-14, vonoprazan (20mg bid) + amoxicillin (1g tid). This regimen combines the staged nature of sequential therapy with the advantages of high-dose dual therapy. The gradual increase in drug dosage may help patients adapt to higher doses while minimizing gastrointestinal discomfort (such as nausea, vomiting, and diarrhea), potentially improving tolerance, especially for those sensitive to antibiotics.

This study aims to evaluate the modified regimen of vonoprazan combined with high-dose amoxicillin in comparison to standard dual therapy (14-day regimen) in terms of HP eradication rates, efficacy, side effect incidence, and patient compliance. Additionally, a multicenter randomized controlled trial in China demonstrated that the 10-day regimen of vonoprazan (20mg bid) + amoxicillin (1g tid) is not inferior to quadruple therapy, with ITT eradication rates of 86% and 89.2%, respectively. Therefore, this study will further explore the impact of shortened treatment duration on the efficacy of the modified dual sequential therapy for HP eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years, gender unrestricted.
2. Chronic gastritis patients with Helicobacter pylori positivity: (1) Helicobacter pylori positive is defined as a positive result on a carbon-13 or carbon-14 breath test within one month prior to enrollment; (2) Chronic gastritis is defined as a diagnosis based on gastroscopy within six months prior to enrollment.
3. No previous Helicobacter pylori eradication therapy.
4. Agree to participate in the trial and sign the informed consent form

Exclusion Criteria:

1. Allergy to any of the drugs used in this clinical trial.
2. Previously received H. pylori eradication treatment.
3. Receiving Potassium-competitive acid blocker (P-CAB), proton pump inhibitor (PPI), H2 receptor antagonist, antibiotics, bismuth, probiotic preparations 4 weeks before initiating study treatment.
4. Use of non-steroidal anti-inflammatory drugs (NSAIDs), adrenal corticosteroids, or anticoagulants during the study period.
5. Pregnant or lactating women, or patients planning to conceive during the study period.
6. Patients with hepatic or renal dysfunction, or those with severe concomitant diseases that may affect the evaluation of this study, such as heart disease, lung disease, liver disease, kidney disease, metabolic disorders, mental illnesses, malignant tumors, etc..
7. Gastroscopy findings indicating conditions other than gastritis, such as reflux esophagitis, which require continued use of potassium-competitive acid blockers (P-CABs), proton pump inhibitors (PPIs), H2 receptor antagonists, or bismuth after Helicobacter pylori eradication.
8. Patients with a history of gastric surgery.
9. Patients who are unable to accurately express their symptoms, such as those with psychiatric disorders or severe neurosis, and are unable to cooperate with the trial.
10. Patients who have participated in other drug studies within 3 months before using the investigational drug.
11. Other conditions deemed by the investigator as unsuitable for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 4-6 weeks after treatment completion
  Rate of H. pylori successfully eradicated; The confirmation of H. pylori status was evaluated by Urea breath test.

SECONDARY OUTCOMES:
Patient compliance | 1 day after treatment completion
  Good compliance was defined as achieving ≥80% of drugs in the regimes and bad compliance was defined as achieving <80% of drugs.
Adverse events | For the 10-day intervention: assessment on Day 5 and Day 10; For the 14-day intervention: assessment on Day 7 and Day 14.
  Adverse drug reactions, including the incidence of both overall and serious adverse events, will be assessed using a standardized questionnaire.
Cost-effectiveness ratio | 1 day after the procedure
  The cost-effectiveness ratio is defined as the total cost per patient for one course of H. pylori eradication treatment divided by the H. pylori eradication rate.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No